CLINICAL TRIAL: NCT04384302
Title: Efficacy of Visual Training in Beach Tennis - a Pilot Study
Brief Title: Efficacy of Visual Training in Beach Tennis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wrocław University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ST001.2020
Record Dates: First submitted 2020-04-17; First posted 2020-05-12 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Visual Performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Visual training (Experimental): Pre-specidied visual training methods that use: the Marsden ball, tables that uses green-red visual stimuli, physical reation in response to the visual stimuli that uses the flippers or the preselected distances.
  One set of exercises per week was prepared.
  Each visual training will last for 15 minutes and should be performed by the participant in their home (using the telemedicine devices to control the conduction of each exercise) 3 times a week.
  Interventions: Other: Visual training

INTERVENTIONS:
Other: Visual training — Pre-defined visual training protocol including the optometrical unit exercises

SUMMARY:
The proposed protocol is going to study the importance of wide spread of visual functions defined by but not limited to visual perception, visual function, visual exploration, involved in the performance of beach tennis. The investigators intend to examine the basic and important visual function that are required for the better performance in the field. The aim is to assess the efficacy of general training that uses the visual channel as the main one. The investigators suspects the improvement in the visual and motor skills after a predefined 8 weeks of visual training.

ELIGIBILITY:
Inclusion Criteria:

* experienced beach tennis player
* participants able and willing to participate in the study (including telemedicine supervision during the training phase)
* known and using full spectacles correction or its equivalent in contact lens correction

Exclusion Criteria:

* inability to give an informed consent
* any disease that causes visual opacity that unable to perform visual training
* participant unable to conduct full visual training course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-05-13 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Optomechanical reaction time | 8 weeks
  The reaction time between the visual stimulus and the motor reaction

SECONDARY OUTCOMES:
Static visual acuity | 8 weeks
  Best-corrected visual acuity in static conditions expressed in logMAR
Dynamic visual acuity | 8 weeks
  Best-corrected visual acuity in dynamic conditions expressed in logMAR
Overall performance during sparing match | 8 weeks
  Overall performance of the player during the supervised match [percentage of properly conducted series of moves specific to rocket sports]

OTHER OUTCOMES:
The pace of macular fixation | 8 weeks
  Checking the pace of macular fixation in the predefined text of equal lenght of words.
Reading rate during the optokinetic task | 8 weeks
  Checking the reading rate during the optokinetic task.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Optics and Photonics, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: No